CLINICAL TRIAL: NCT03062176
Title: Interleukin-1 Blockade for the Treatment of Heart Failure in Patients With Advanced Chronic Kidney Disease (E-HART)
Brief Title: Interleukin-1 Blockade for the Treatment of Heart Failure in Patients With Advanced Chronic Kidney Disease
Acronym: E-HART
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: We screened over 200 patients but were ultimately unable to enroll anyone
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM20007618
Record Dates: First submitted 2017-01-25; First posted 2017-02-23 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Heart Failure, Systolic; Renal Disease, End Stage; Chronic Kidney Diseases
Keywords: Heart failure; End-stage renal disease; Interleukin-1; Interleukin-1 receptor antagonist; Metabolomics; Lipidomics; Chronic kidney disease
MeSH Terms: conditions — Heart Failure, Systolic; Kidney Failure, Chronic; Renal Insufficiency, Chronic; Heart Failure | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Active Treatment (Experimental): Anakinra (Kineret)
  Interventions: Drug: Anakinra

INTERVENTIONS:
Drug: Anakinra — Anakinra (Kineret)
  Other Names: Kineret

SUMMARY:
Interleukin-1 blockade for the treatment of heart failure in patients with advanced chronic kidney disease (End-stage renal disease and Heart fAilure - Anakinra Remodeling Trial) is a Phase 2, single-arm trial designed to estimate the effect of anakinra, a recombinant human Interleukin-1 (IL-1) receptor antagonist, on cardiorespiratory fitness in patients with advanced chronic kidney disease and heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* 18 years or older
* Chronic heart failure
* Left ventricular ejection fraction less than 50%
* C-reactive protein greater than or equal to 2 mg/L
* Maintenance hemodialysis with a biocompatible membrane, acceptable dialysis adequacy (Kt/V > 1.2), and receipt of a stable hemodialysis prescription for at least 4 weeks OR chronic kidney disease stage IV/V (estimated glomerular filtration rate <30 mL/min/1.73m2)

Exclusion Criteria:

* Inability to complete maximal cardiopulmonary exercise testing
* Need for urgent or emergent care
* Recent use of immunosuppressant, anti-inflammatory therapies or active rheumatologic disease
* Allergy to rubber, latex, Escherichia coli or anakinra

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Peak oxygen consumption (PVO2) | 6 months
  Peak oxygen consumption during cardiopulmonary exercise

SECONDARY OUTCOMES:
Heart Failure Hospitalization | 6 months
  Number of participants with a hospitalization for heart failure during the 6 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin W Van Tassell, PharmD, Principal Investigator — Virginia Commonwealth University